CLINICAL TRIAL: NCT02200159
Title: Predictive Factors of Failure or Success of Sedation With Dexmedetomidine in ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0197; 2013-000960-26
Record Dates: First submitted 2014-06-30; First posted 2014-07-25 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Requiring Sedation in ICU; Adult Patients; Patient Covered by French Health Care System
Keywords: Sedation; Dexmedetomidine; ICU; Delirium
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (1):
- dexmedetomidine
  Interventions: Drug: Sedation with dexmedetomidine

INTERVENTIONS:
Drug: Sedation with dexmedetomidine

SUMMARY:
Research predictive factors of success or failure of a sedation with Dexmedetomidine in ICU

DETAILED DESCRIPTION:
Prospective clinical study in ICU with sedated ventilated patients with dexmedetomidine, establishing incidence of success, failure of moderate sedation or failure of dexmedetomidine, to evaluate the effectiveness of this drug sedation in moderate sedation

ELIGIBILITY:
Inclusion Criteria:

-Adult patients ventilated requiring sedation in ICU with RASS objective more than -2

Exclusion Criteria:

* contraindication: intracranial lesion, hepatic failure
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients ventilated requiring sedation in ICU with RASS objective more than -2
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with failure of sedation with dexmedetomidine | at day 1
  Number of patients with failure of sedation with dexmedetomidine (necessity to stop this sedation due to adverse event, RASS>+1, other) in ICU patients requiring such sedation during ICU stay.

SECONDARY OUTCOMES:
Incidence of adverse event of dexmedetomidine | at day 1
Incidence of delirium and use of other sedative drugs | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel CONSTANTIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France